CLINICAL TRIAL: NCT05318170
Title: Evaluation of Surgical Outcomes After Laparoscopic Ultra-radical Lymph Node Debulking Using Yasargil Clamps for Gynecological Malignancies
Brief Title: Laparoscopic Ultra-radical Lymph Node Debulking Using Yasargil Clamps (Yasargil-1)
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Collaborators: Fondazione Policlinico Universitario A. Gemelli, IRCCS (Unknown); Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, University of Palermo
Other Study IDs: Yasargil-1
Record Dates: First submitted 2022-04-04; First posted 2022-04-08 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Gynecologic Cancer
Keywords: Gynecological oncology; Gynecological cancers; Bulky lymph nodes; Laparoscopic ultra-radical lymph node debulking; Yasargil clamps; Complications; Surgical outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women affected by gynecological cancer: Women affected by gynecological cancer (cervical, endometrial, ovarian and vulvar cancer)
  Interventions: Procedure: Laparoscopic ultra-radical lymph node debulking

INTERVENTIONS:
Procedure: Laparoscopic ultra-radical lymph node debulking — Laparoscopic ultra-radical lymph node debulking using Yasargil clamps

SUMMARY:
Although several studies have demonstrated the overall benefits of a laparoscopic approach for pelvic and para-aortic lymphadenectomy, complications remain a challenging scenario. Vascular injury occurs in 0.3% to 1.0% of laparoscopic procedures, with potentially lethal consequences. Vascular injuries are usually managed using coagulation, clamps or vascular sutures, but if these measures fail, laparotomy is inevitable.

To date, few reports evaluated the use of minimally invasive surgery for lymph node debulking in gynecological cancer patients with metastatic bulky lymph nodes, with encouraging results, despite the small sample sizes. Nevertheless, new minimally invasive surgery techniques that may minimize intraoperative complications are necessary. Considering these elements, this multicenter retrospective analysis is aimed to evaluate intra- and post-operative surgical outcomes, after laparoscopic ultraradical lymph nodal debulking using Yasargil clamps in gynecological cancer patients with bulky lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* At least one bulky lymph node with size ≥ 25 mm
* Age > 18 years
* Body mass index (BMI) < 40 kg/m²
* Absence of abdominal adhesion syndrome and intraperitoneal dissemination at the time of laparoscopic evaluation

Exclusion Criteria:

* Disease-free interval < 6 months and/or
* Performance status > 2 according to Eastern Cooperative Oncology Group (ECOG) criteria

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women affected by gynecological cancer.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Complications | During the surgery and within 30 days after the surgery
  Any complication occurred

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Study Chair — University of Palermo; Vito Chiantera, Study Director — University of Palermo; Mariano Catello Di Donna, Principal Investigator — University of Palermo
Locations (1):
- University of Palermo, Palermo, Sicily, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Donna MC, Sozzi G, Cucinella G, Giallombardo V, Gallotta V, Uccella S, Garzon S, Scambia G, Lagana AS, Chiantera V. Laparoscopic Ultra-radical Lymph Node Debulking Using Yasargil Clamps for Gynecological Malignancies: Results from a Large, Multicenter, Retrospective Analysis. J Minim Invasive Gynecol. 2022 Sep;29(9):1083-1091. doi: 10.1016/j.jmig.2022.05.016. Epub 2022 May 29. PMID 35649479